CLINICAL TRIAL: NCT02528630
Title: Effectiveness of a Progressive Resistance Strength Program on Hand Osteoarthritis: a Randomized Controlled Trial
Brief Title: Progressive Strength in Hand Osteoarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Michele Nery, Master Student, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEP UNIFESP
Record Dates: First submitted 2015-08-17; First posted 2015-08-19 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Hand Osteoarthritis

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Exercise group (Experimental): Performed a session regarding joint protection and energy conservation and a progressive resistance strength training program for intrinsic muscles of the hand for 12 weeks.
  Interventions: Other: Progressive resistance strength training program; Other: Joint protection and energy conservation advice
- Control group (Active Comparator): Performed a session regarding joint protection and energy conservation
  Interventions: Other: Joint protection and energy conservation advice

INTERVENTIONS:
Other: Progressive resistance strength training program — Patients undergo to strength training for intrinsic muscles of the hand twice a week, during 12 weeks.
  Arms: Exercise group
Other: Joint protection and energy conservation advice — A session regarding joint protection and energy conservation for hands was done before randomization.

SUMMARY:
Background: Hand osteoarthritis (OA) is highly prevalent, affecting 55-70% of the population over 55 years with an age-related progressive increase. The OA of interphalangeal (IF) and carpometacarpal joints may have varying degrees of deformity associated with pain, decreased of grip and pinch strength, decreased range of motion and functional impairment. Systematic reviews and meta-analyzes have shown the beneficial effect of exercise for lower limb OA, however for hand OA exercise is still used based on recommendations based on clinical experience and low quality studies, not allowing a conclusion about the effects of exercise in pain, function and strength in hand OA patients.

Objective: assess the effectiveness of progressive resistance strength training program on pain, function and strength in hand OA patients.

Methods: diagnostic of hand OA according to American College of Rheumatology of at least 1year, age over 50 years, both genders, pain in IF joints between 3-8 cm on a 10-cm numerical pain scale (NPS). Sixty patients who meet the eligibility criteria were randomized into exercise group (EG) and control group (CG). Both groups performed a session regarding joint protection and energy conservation before randomization. The EG performed a progressive resistance strength training program for intrinsic muscles of the hand for 12 weeks. The outcome measures were NPS; Australian/Canadian (AUSCAN) Hand Osteoarthritis Index and Cochin Hand Functional Scale for hand function; grip and pinch strengthening using the Hydraulic Hand Dynamometer and a pinch gauge dynamometer and satisfaction with the treatment using a Likert scale. A blinded evaluator performed the evaluations at baseline, 6 and 12 weeks after treatment baseline.

ELIGIBILITY:
Inclusion Criteria:

* diagnostic of hand OA according to american college of rheumatology of at least 1year;
* age over 50 years;
* both genders;
* pain in interphalangeal joints between 3-8 cm on a 10-cm numerical pain scale

Exclusion Criteria:

* other joint disease in hands;
* other rheumatic systemic disease;
* surgery in hands or writs;
* exercise or joint injection in hands in the previous 3 months;
* disability to perform the exercises.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-10; Primary Completion 2015-01 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in Pain | Baseline, after 6 and 12 weeks
  Measured by a numerical pain scale

SECONDARY OUTCOMES:
Change in hand function | Baseline, after 6 and 12 weeks
  measured by AUSCAN
Change in Patient satisfaction with treatment | 6 and 12 weeks
  Measured by a Likert scale
Change in grip strength | Baseline, after 6 and 12 weeks
  Measured by a Grip Hydraulic Hand Dynamometer
Change in hand function | Baseline, after 6 and 12 weeks
  Measured by COCHIN questionnaires
Change in pinch stength | Baseline, after 6 and 12 weeks
  Measured by pinch gauge dynamometer

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de Sao Paulo, São Paulo, São Paulo, Brazil